CLINICAL TRIAL: NCT05071742
Title: Correlation of Genetic Susceptibility Genes to Inflammatory Bowel Disease in Chinese Han Population
Acronym: CGSGIBDCHP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiao xiao Shao, attending doctor, Second Affiliated Hospital of Wenzhou Medical University
Other Study IDs: SAHoWMU-CR2021-01-206
Record Dates: First submitted 2021-09-24; First posted 2021-10-08 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Gene Abnormality; Inflammatory Bowel Disease; Chinese
Keywords: IBD;gene;Chinese Han population
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole-genome DNA extraction: 2 mL peripheral fasting venous blood was extracted from IBD patients or control group, and edTA disodium was anticoagulant.The whole genome DNA was extracted in strict accordance with the instructions of the blood genomic DNA extraction Kit. The concentration and purity of DNA were detected by nanodrop-1000 spectrophotometer. The DNA was diluted to 10 ng/μL and stored in the refrigerator at -80℃ for future use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD group: According to the consensus opinions on diagnosis and Treatment of Inflammatory Bowel Disease (Beijing, 2018) formulated by Chinese Society of Gastroenterology, Chinese Medical Association The diagnosis of IBD was confirmed by clinical, laboratory, radiographic, digestive endoscopy and histopathological examination.
  Interventions: Genetic: 2ml peripheral venous blood was collected to detect genetic genes
- control group: During the same period, healthy subjects were collected from the physical examination center of our hospital as subjects of the normal control group. Infectious diarrhea, ischemic bowel disease, radiation enteritis, gastrointestinal tumor, diabetes, systemic lupus erythematosus, rheumatoid arthritis and autoimmune thyroiditis were excluded from all clinical examinations before inclusion.
  Interventions: Genetic: 2ml peripheral venous blood was collected to detect genetic genes

INTERVENTIONS:
Genetic: 2ml peripheral venous blood was collected to detect genetic genes — Extraction of whole genome DNA: 2 mL of peripheral fasting venous blood was extracted, and edTA disodium was anticoagulant.The whole-genome DNA was extracted strictly in accordance with the instructions of the blood genomic DNA extraction kit (Beijing Tiagen Biochemical Technology Co., LTD., China), and the DNA concentration and purity were detected by nanodrop-1000 spectrophotometer (Thermo, USA). The DNA was diluted to 10 ng/μL and stored in a refrigerator at -80℃ for future use.
  (2) Primer design and synthesis: (3) Gene polymorphism detection 4) Resin purification 5) Spot chip and mass spectrometry detection
  Other Names: DNA is extracted and genetic testing is performed

SUMMARY:
The pathogenesis of IBD is still unclear, and the disease characteristics of IBD patients are affected by genetic susceptibility genes. Therefore, this study aims to explore the relationship between genetic susceptibility genes of IBD and the pathogenesis of IBD in Chinese Han population, in order to clarify the pathogenesis of IBD and provide basis for individualized treatment of IBD.

DETAILED DESCRIPTION:
The pathogenesis of IBD is still unclear, and the disease characteristics of IBD patients are affected by genetic susceptibility genes. Therefore, this study aims to explore the relationship between genetic susceptibility genes of IBD and the pathogenesis of IBD in Han Chinese, in order to clarify the pathogenesis of IBD and provide basis for individualized treatment of IBD.In this study, 5ml peripheral venous blood was drawn from IBD patients and normal controls for gene testing.To investigate the relationship between polymorphisms of TRAIL, ITGA4, ICAM1, ITGA4, ICAM1, LTA, FCGR3A, TRAP1, TNFRSF1B, CDKN2B-AS1 and susceptibility to IBD in Chinese Han population.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed IBD patients were collected from the Department of Gastroenterology, The Second Affiliated Hospital of Wenzhou Medical University.According to the consensus of "Diagnosis and treatment of inflammatory bowel disease" formulated by Chinese Society of Gastroenterology, the diagnosis of IBD was established by clinical, laboratory, radiographic, digestive endoscopy and histopathological examination.During the same period, 476 healthy subjects were collected from the physical examination center of our hospital as the normal control group

Exclusion Criteria:

* Active infection, malignant tumor, congestive heart failure, demyelination of nervous system, allergy to rat derived protein components, etc All subjects were excluded from infectious diarrhea, ischemic enteropathy, radiation enteritis, gastrointestinal tumor, diabetes, systemic lupus erythematosus, rheumatoid arthritis and autoimmune thyroiditis by clinical examination before inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Adults who have not undergone acquired sex reassignment surgery can be included
Study Population: IBD patients or healthy controls who met the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-11-25 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of genetic susceptibility genes to inflammatory bowel disease in Chinese Han population | 2021-2024
  The difference in mutation frequency of different gene loci between IBD patients and control group was compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Li, PHD, Study Director — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No